CLINICAL TRIAL: NCT07114341
Title: Effect of Lyophilized Cornelian Cherry on Anaerobic Performance in Young Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Hande Seven Avuk, Assistant Professor, Head of Nutrition and Dietetic Department, Istanbul Bilgi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CORNELIANCHERRYFOOTBALLSTUDY
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Sport Nutrition; Sports Performance in Children; Ergogenic Athletic Performance; Ergogenic Support; Sports Nutritional Sciences
Keywords: cranberry; sports nutrition; ergogenic acids; football; adolecent athletes

STUDY DESIGN:
Intervention Model Description: This study designed as an intervention study.
Masking Description: Not suitable for masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): In order to determine the standard performance of the adolescent football players in the first stage before the intervention, a Running-Based Anaerobic Sprint Test (RAST) was applied to the adolescent football players on a grass field in an open-air environment after a 10-minute warm-up exercise.
- Cranberry Intervention (Active Comparator): In the second phase of the study, adolescent soccer players were given 30 grams of freeze-dried cranberries containing 1187 mg/100 g anthocyanins daily for 1 week. To determine post-intervention performance, the adolescent soccer players underwent a 10-minute warm-up exercise followed by a Running-Based Anaerobic Sprint Test (RAST) on a grass field in an outdoor environment.
  Interventions: Other: Cranberry Intervention

INTERVENTIONS:
Other: Cranberry Intervention — 30 grams of lyophilized cranberry containing 1187 mg/100 g anthocyanins were given for 7 days.
  Arms: Cranberry Intervention

SUMMARY:
The goal of this clinical trial is to learn if a lyophilized Cornelian Cherry supplement works to improve anaerobic performance and reduce fatigue in young football players (U14-U19 age group).

The main questions it aims to answer are:

* Does taking a lyophilized Cornelian Cherry supplement improve participants' anaerobic performance as measured by the Running-based Anaerobic Sprint Test (RAST)?
* Does the supplement reduce participants' levels of fatigue after strenuous exercise?

Researchers will measure participants' performance and fatigue levels before the study begins and compare them to the levels measured after 1 week of taking the cranberry supplement. This will help determine the effect of the supplement.

Participants will:

* Take 30 grams of lyophilized Cornelian Cherry powder every day for 1 week.
* Visit the study center at the beginning and at the end of the 1-week period for checkups and tests.
* Undergo anthropometric measurements (such as height, weight, and body composition) at the start of the study.
* Perform a Running-based Anaerobic Sprint Test (RAST) and a fatigue test at the start and end of the study.

DETAILED DESCRIPTION:
A balanced diet plays a role in preventing injuries, improving athletic performance, and accelerating post-exercise recovery in adolescents who engage in physical activity. The physiological response to exercise can vary depending on the duration, intensity, and frequency of exercise, as well as environmental conditions. Excessive reactive oxygen species (ROS) production triggered by high-intensity exercise or other stress factors in athletes can lead to oxidative stress and subsequent tissue damage by weakening the antioxidant defense system. Therefore, athletes may need to maintain increased ROS scavenging activity. Additionally, physical exercise can lead to injuries in skeletal muscle tissue, leading to decreased performance. Therefore, strategies to manage exercise-related injuries and post-exercise inflammatory processes may contribute to accelerating exercise adaptation and recovery. Recently, there has been increasing support for the possibility of improving exercise performance through supplementation with fruit-derived polyphenols. Polyphenols are secondary metabolites abundant in plant foods and are divided into four main groups: lignans, stilbenes, and flavonoids. Anthocyanins, a subclass of flavonoids, are found in red, purple, and blue vegetables and fruits. Anthocyanins are known for their antioxidant and anti-inflammatory properties, and therefore, they are thought to prevent adverse physiological effects such as fatigue and post-exercise inflammation, which can potentially occur during exercise. The potential mechanism of action is thought to be related to antioxidant and vascular effects. Turkey is among the countries where cornelian cherries, another fruit with high biological value due to their anthocyanin and other phenolic compounds, are cultivated. Randomized controlled trials have examined the effectiveness of freeze-dried cornelian cherry supplements in various disease groups. Studies have observed positive effects on lipid profiles, as well as parameters related to body mass index (BMI), body weight, waist and hip circumference, and insulin resistance. Another randomized controlled trial has indicated that cornelian cherry supplementation may be effective in accelerating post-exercise recovery in athletes. While the literature has evaluated the effects of various forms of supplementation with fruits high in anthocyanins on sports performance, studies examining anaerobic power and capacity with cornelian cherry supplementation in adolescent athletes are limited. Therefore, the purpose of this study was to evaluate the effects of freeze-dried cornelian cherry fruit on anaerobic performance in adolescent soccer players.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 ages of adolescent football

Exclusion Criteria:

* Disease diagnosis or history,
* Regular medication use,
* Regular nutritional supplement use,
* Being under 14 years of age,
* Being over 19 years of age.

Ages: 14 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Running-Based Anaerobic Sprint Test (RAST) - Performance Test | From enrollment to the end of study at 1 week
  The RAST is a test consisting of six 35-meter sprints at maximum speed, with a 10-second rest interval between each sprint. In this test, power is calculated for each sprint using body mass and the resulting performance data (Power = (Total body mass x Distance2) / Time3). The highest recorded number is called maximum power; the lowest number is called minimum power; and the sum of the six sprints divided by six is called average power. Muscle fatigue is assessed using the Fatigue Index (Maximum Power - Minimum Power) / Sum of the 6 sprint times). A lower value indicates that athletes have better muscular ability to maintain their performance without fatigue.

SECONDARY OUTCOMES:
Anthropometric Measurements - Body weight (kg) | From enrollment to the end of study at 1 week
  At the beginning and end of the study, body weights (kg) measured using a bioelectrical impedance (BIA) device with a sensitivity of 50 grams in accordance with the measurement standards.
Anthropometric Measurements - Height | 1 week
  Height (cm) measured with a stadiometer in the Frankfort plane, standing and with the head upright.
Body Mass Index | From enrollment to the end of study at 1 week
  The body mass index (BMI) of the participants was calculated according to the body weight (kg) / height (m)2 formula.
Anthropometric Measurements - Fat Mass | From enrollment to the end of study at 1 week
  At the beginning and end of the study, body fat mass (kg) analysis was performed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Fat ratio calculation | From enrollment to the end of study at 1 week
  At the beginning and end of the study, body composition analyses was performed using a bioelectrical impedance (BIA) device with measurement standards. According to the BIA analysis, fat percentage (%) will be calculated as the ratio of total body fat weight to total body weight.
Anthropometric Measurements - Fat-free mass | From enrollment to the end of study at 1 week
  At the beginning and end of the study, fat-free mass (kg) was analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Muscle mass | From enrollment to the end of study at 1 week
  At the beginning and end of the study, lean muscle mass (kg) was analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Anthropometric Measurements - Total body water | From enrollment to the end of study at 1 week
  At the beginning and end of the study, total body water (kg) was analyzed using a bioelectrical impedance (BIA) device, paying attention to measurement standards.
Food Consumption Record - Energy | 1 day
  The food consumption record was taken to evaluate the nutritional status of the participants. Food consumption records were evaluated in the BeBIS (Nutrition Information System) program and the daily energy (kcal) intake will be calculated.
Food Consumption Record | 1 day
  The food consumption record were taken to evaluate the nutritional status of the participants. Food consumption records were evaluated in the BeBIS (Nutrition Information System) program and the daily carbohydrate (g), protein (g), fat (g), saturated fat (g), monounsaturated fatty acid (g), polyunsaturated fatty acid (g), omega-3 fatty acids (g), omega-6 fatty acids (g), and fiber (g) intake were calculated.
Food Consumption Record | 1 day
  The food consumption record was taken to evaluate the nutritional status of the participants. Food consumption records were evaluated in the BeBIS (Nutrition Information System) program and the daily vitamin A (µg), vitamin D (µg), vitamin K (µg), folate (µg), and vitamin B12 (µg) intake were calculated.
Food Consumption Record | 1 day
  The food consumption record was taken to evaluate the nutritional status of the participants. Food consumption records were evaluated in the BeBIS (Nutrition Information System) program and the daily vitamin E (mg), thiamine (mg), riboflavine (mg), niacin (mg), vitamine B5 (mg), vitamin B6 (mg), vitamin C, sodium (mg), potassium (mg), calcium (mg), magnesium (mg), phosphor (mg), iron (mg), zinc (mg), copper (mg), cholesterol (mg) intake were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braakhuis AJ, Somerville VX, Hurst RD. The effect of New Zealand blackcurrant on sport performance and related biomarkers: a systematic review and meta-analysis. J Int Soc Sports Nutr. 2020 May 27;17(1):25. doi: 10.1186/s12970-020-00354-9. PMID 32460873
- [Background] Donno D, Neirotti G, Fioccardi A, Razafindrakoto ZR, Tombozara N, Mellano MG, Beccaro GL, Gamba G. Freeze-Drying for the Reduction of Fruit and Vegetable Chain Losses: A Sustainable Solution to Produce Potential Health-Promoting Food Applications. Plants (Basel). 2025 Jan 9;14(2):168. doi: 10.3390/plants14020168. PMID 39861522
- [Background] Jastrzebska AD. Comparison of usefulness of two tests measuring anaerobic performance of untrained and soccer-training girls U12. Sci Rep. 2023 Nov 9;13(1):19498. doi: 10.1038/s41598-023-46825-2. PMID 37945713
- [Background] Rizal M, Segalita C, Mahmudiono T. The Relationship between Body Mass Index, Body Fat Percentage, and Dietary Intake with Muscle Fatigue in Adolescent Football Players. J Nutr Sci Vitaminol (Tokyo). 2020;66(Supplement):S134-S136. doi: 10.3177/jnsv.66.S134. PMID 33612582
- [Background] Bayram HM, Iliaz R, Gunes FE. Effects of Cornus mas L. on anthropometric and biochemical parameters among metabolic associated fatty liver disease patients: Randomized clinical trial. J Ethnopharmacol. 2024 Jan 10;318(Pt B):117068. doi: 10.1016/j.jep.2023.117068. Epub 2023 Aug 21. PMID 37611681
- [Background] Kazimierski M, Regula J, Molska M. Cornelian cherry (Cornus mas L.) - characteristics, nutritional and pro-health properties. Acta Sci Pol Technol Aliment. 2019 Jan-Mar;18(1):5-12. doi: 10.17306/J.AFS.0628. PMID 30927747
- [Background] Godwin C, Cook MD, Willems MET. Effect of New Zealand Blackcurrant Extract on Performance during the Running Based Anaerobic Sprint Test in Trained Youth and Recreationally Active Male Football Players. Sports (Basel). 2017 Sep 15;5(3):69. doi: 10.3390/sports5030069. PMID 29910429
- [Background] Khoo HE, Azlan A, Tang ST, Lim SM. Anthocyanidins and anthocyanins: colored pigments as food, pharmaceutical ingredients, and the potential health benefits. Food Nutr Res. 2017 Aug 13;61(1):1361779. doi: 10.1080/16546628.2017.1361779. eCollection 2017. PMID 28970777
- [Background] Bowtell J, Kelly V. Fruit-Derived Polyphenol Supplementation for Athlete Recovery and Performance. Sports Med. 2019 Feb;49(Suppl 1):3-23. doi: 10.1007/s40279-018-0998-x. PMID 30671906
- [Background] Bolat E, Saritas S, Duman H, Eker F, Akdasci E, Karav S, Witkowska AM. Polyphenols: Secondary Metabolites with a Biological Impression. Nutrients. 2024 Aug 3;16(15):2550. doi: 10.3390/nu16152550. PMID 39125431
- [Background] Volpe-Fix AR, de Franca E, Silvestre JC, Thomatieli-Santos RV. The Use of Some Polyphenols in the Modulation of Muscle Damage and Inflammation Induced by Physical Exercise: A Review. Foods. 2023 Feb 21;12(5):916. doi: 10.3390/foods12050916. PMID 36900433
- [Background] Sawada Y, Ichikawa H, Ebine N, Minamiyama Y, Alharbi AAD, Iwamoto N, Fukuoka Y. Effects of High-Intensity Anaerobic Exercise on the Scavenging Activity of Various Reactive Oxygen Species and Free Radicals in Athletes. Nutrients. 2023 Jan 1;15(1):222. doi: 10.3390/nu15010222. PMID 36615878
- [Background] He F, Li J, Liu Z, Chuang CC, Yang W, Zuo L. Redox Mechanism of Reactive Oxygen Species in Exercise. Front Physiol. 2016 Nov 7;7:486. doi: 10.3389/fphys.2016.00486. eCollection 2016. PMID 27872595
- [Background] Capra ME, Stanyevic B, Giudice A, Monopoli D, Decarolis NM, Esposito S, Biasucci G. Nutrition for Children and Adolescents Who Practice Sport: A Narrative Review. Nutrients. 2024 Aug 22;16(16):2803. doi: 10.3390/nu16162803. PMID 39203939
- [Background] Amawi A, Khataybeh B, Al Aqaili R, Ababneh N, Alnimer L, Qoqazeh A, Oukal F, Jahrami H, Mousa Ay K, Al Saoud H, Ghazzawi H. Junior athletes' nutritional demands: a narrative review of consumption and prevalence of eating disorders. Front Nutr. 2024 Sep 24;11:1390204. doi: 10.3389/fnut.2024.1390204. eCollection 2024. PMID 39381351